CLINICAL TRIAL: NCT03001076
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of Bempedoic Acid (ETC 1002) 180 mg/Day as Add-on to Ezetimibe Therapy in Patients With Elevated LDL-C
Brief Title: Evaluation of the Efficacy and Safety of Bempedoic Acid (ETC-1002) as Add-on to Ezetimibe Therapy in Patients With Elevated LDL-C (CLEAR Tranquility)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1002-048
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesterolemia; Atherosclerosis; Statin Adverse Reaction
Keywords: hyperlididemia; LDL; cholesterol; statin intolerance
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bempedoic acid (Experimental): bempedoic acid 180 mg tablet taken orally, daily. Patients remain on ongoing ezetimibe therapy (study provided)
  Interventions: Drug: Bempedoic acid; Drug: Ezetimibe
- placebo (Placebo Comparator): Matching placebo tablet taken orally, daily. Patients remain on ongoing ezetimibe therapy (study provided)
  Interventions: Drug: Ezetimibe; Other: Placebo

INTERVENTIONS:
Drug: Bempedoic acid — bempedoic acid 180 mg tablet
  Other Names: ETC-1002
  Arms: bempedoic acid
Drug: Ezetimibe — ezetimibe 10 mg tablet
  Other Names: Zetia
Other: Placebo — matching placebo tablet
  Other Names: placebo control
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if bempedoic acid (ETC-1002) added-on to ezetimibe therapy is effective and safe versus placebo in patients with elevated LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Fasting LDL-cholesterol greater than or equal to 100 mg/dL at screening
* Men and nonpregnant, nonlactating women
* Use of stable lipid-modifying therapy for at least 4 weeks prior to screening that includes ezetimibe 10mg daily

Exclusion Criteria:

* Fasting blood triglycerides greater than or equal to 500 mg/dL
* Body Mass Index (BMI) greater than or equal to 50 kg/m2
* Recent history of clinically significant cardiovascular disease
* Use of statin therapy where doses are greater than those defined as "low-dose" within 4 weeks prior to screening; where "low-dose" is defined as an average daily dose of rosuvastatin 5 mg, atorvastatin 10 mg, simvastatin 10 mg, lovastatin 20 mg, pravastatin 40 mg, fluvastatin 40 mg, or pitavastatin 2 mg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Haberman, MD, Study Director — Esperion Therapeutics, Inc.
Locations (1):
- Georgetown, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinkosky SL, Newton RS, Day EA, Ford RJ, Lhotak S, Austin RC, Birch CM, Smith BK, Filippov S, Groot PHE, Steinberg GR, Lalwani ND. Liver-specific ATP-citrate lyase inhibition by bempedoic acid decreases LDL-C and attenuates atherosclerosis. Nat Commun. 2016 Nov 28;7:13457. doi: 10.1038/ncomms13457. PMID 27892461
- [Background] Bilen O, Ballantyne CM. Bempedoic Acid (ETC-1002): an Investigational Inhibitor of ATP Citrate Lyase. Curr Atheroscler Rep. 2016 Oct;18(10):61. doi: 10.1007/s11883-016-0611-4. PMID 27663902
- [Background] Thompson PD, MacDougall DE, Newton RS, Margulies JR, Hanselman JC, Orloff DG, McKenney JM, Ballantyne CM. Treatment with ETC-1002 alone and in combination with ezetimibe lowers LDL cholesterol in hypercholesterolemic patients with or without statin intolerance. J Clin Lipidol. 2016 May-Jun;10(3):556-67. doi: 10.1016/j.jacl.2015.12.025. Epub 2016 Jan 6. PMID 27206943
- [Background] Ballantyne CM, McKenney JM, MacDougall DE, Margulies JR, Robinson PL, Hanselman JC, Lalwani ND. Effect of ETC-1002 on Serum Low-Density Lipoprotein Cholesterol in Hypercholesterolemic Patients Receiving Statin Therapy. Am J Cardiol. 2016 Jun 15;117(12):1928-33. doi: 10.1016/j.amjcard.2016.03.043. Epub 2016 Apr 6. PMID 27138185
- [Background] Thompson PD, Rubino J, Janik MJ, MacDougall DE, McBride SJ, Margulies JR, Newton RS. Use of ETC-1002 to treat hypercholesterolemia in patients with statin intolerance. J Clin Lipidol. 2015 May-Jun;9(3):295-304. doi: 10.1016/j.jacl.2015.03.003. Epub 2015 Mar 19. PMID 26073387
- [Result] Ballantyne CM, Banach M, Mancini GBJ, Lepor NE, Hanselman JC, Zhao X, Leiter LA. Efficacy and safety of bempedoic acid added to ezetimibe in statin-intolerant patients with hypercholesterolemia: A randomized, placebo-controlled study. Atherosclerosis. 2018 Oct;277:195-203. doi: 10.1016/j.atherosclerosis.2018.06.002. Epub 2018 Jun 12. PMID 29910030
- [Derived] Ballantyne CM, Bays HE, Louie MJ, Smart J, Zhang Y, Ray KK. Factors Associated With Enhanced Low-Density Lipoprotein Cholesterol Lowering With Bempedoic Acid. J Am Heart Assoc. 2022 Aug 2;11(15):e024531. doi: 10.1161/JAHA.121.024531. Epub 2022 Aug 2. PMID 35916348
- [Derived] Banach M, Duell PB, Gotto AM Jr, Laufs U, Leiter LA, Mancini GBJ, Ray KK, Flaim J, Ye Z, Catapano AL. Association of Bempedoic Acid Administration With Atherogenic Lipid Levels in Phase 3 Randomized Clinical Trials of Patients With Hypercholesterolemia. JAMA Cardiol. 2020 Oct 1;5(10):1124-1135. doi: 10.1001/jamacardio.2020.2314. PMID 32609313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of the 269 participants who were randomized to the double-blind treatment period, 181 participants were randomized to bempedoic acid and 88 participants to placebo. One participant in the placebo group was randomized but never started treatment.
Pre-assignment Details: The study consisted of an approximate 1-week screening period, a 4-week single-blind placebo and ezetimibe run-in period, and a 12-week double-blind treatment period.
Groups:
- Placebo: Participants received placebo tablet, once-daily by mouth and ezetimibe 10 mg capsules, once-daily by mouth for 4 weeks prior to the 12-week treatment period. During the treatment period, participants received placebo tablet, once-daily by mouth and ezetimibe 10 mg capsules, once-daily by mouth for 12 weeks.
- Bempedoic Acid: Participants received placebo tablet, once-daily by mouth and ezetimibe 10 mg capsules, once-daily by mouth for 4 weeks prior to the 12-week treatment period. During the treatment period, participants received bempedoic acid 180 mg tablet, once-daily by mouth and ezetimibe 10 mg capsules, once-daily by mouth for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Bempedoic Acid
Started | 88 | 181
Completed | 81 | 176
Not Completed | 7 | 5
Not completed — Withdrawal by patient | 2 | 0
Not completed — Other | 1 | 0
Not completed — Adverse Event | 3 | 3
Not completed — Sponsor decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bempedoic Acid | Total
Number analyzed (Participants) | 88 | 181 | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (11.32) | 63.8 (10.77) | 63.8 (10.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 109 | 165
  Male | 32 | 72 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 43 | 66
  Not Hispanic or Latino | 65 | 138 | 203
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 10 | 11 | 21
  White | 75 | 165 | 240
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
LDL-C category [Count of Participants; unit: Participants]
  <130 mg/dL | 56 | 99 | 155
  ≥130 to <160 mg/dL | 24 | 53 | 77
  ≥160 mg/dL | 8 | 29 | 37
Concomitant lipid-modifying therapy medications [Count of Participants; unit: Participants] — Concomitant medications were defined as medications that started prior to, on or after the first dose of double-blind IMP and started no later than 30 days following end of double-blind IMP, and ended on or after the date of first dose of double-blind IMP or were ongoing at the end of the study. Other LMT included fish oil, eicosapentaenoic acid ethyl ester, omega-3 fatty acids, salmon oil, and sitosterol. Participants received ezetimibe 10 mg/day as background therapy throughout the study. Participants who took at least one concomitant LMT have been reported.
  Participants
    Statins | 25 | 59 | 84
    Fibrates | 3 | 7 | 10
    Nicotinic acid and derivatives | 4 | 3 | 7
    Bile acid sequestrants | 1 | 1 | 2
    Other lipid-modifying therapies | 8 | 19 | 27
    No concomitant lipid-modifying therapies | 47 | 92 | 139
Concomitant illness: Cardiac disorder [Count of Participants; unit: Participants] — Concomitant illness was defined as the present condition that started prior to the date of randomization and was ongoing at the time of randomization.
  Participants
    Participants with cardiac disorder | 22 | 49 | 71
    Participants without cardiac disorder | 66 | 132 | 198
History of diabetes [Count of Participants; unit: Participants]
  Participants with history of diabetes | 17 | 35 | 52
  Participants without history of diabetes | 71 | 146 | 217
History of hypertension [Count of Participants; unit: Participants]
  Participants with history of hypertension | 51 | 111 | 162
  Participants without history of hypertension | 37 | 70 | 107
Estimated glomerular filtration rate (eGFR) category [Count of Participants; unit: Participants] — milliliter per minutes per 1.73 square meter (mL/min/1.73m2)
  Participants
    ≥90 mL/min/1.73m2 | 17 | 45 | 62
    60 to <90 mL/min/1.73m2 | 57 | 110 | 167
    <60 mL/min/1.73m2 | 14 | 26 | 40
Low-density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline was defined as the mean of the last two non-missing values on or prior to Day 1.
  milligrams per deciliter (mg/dL) | 123.02 (27.197) | 129.77 (30.871) | 127.56 (29.838)
Non-high-density lipoprotein cholesterol (non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the last two non-missing values on or prior to Day 1.
  mg/dL | 151.55 (32.734) | 162.41 (35.413) | 158.85 (34.874)
Total cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the last two non-missing values on or prior to Day 1.
  mg/dL | 208.62 (35.712) | 218.24 (35.883) | 215.09 (36.045)
Apolipoprotein B (apoB) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the last non-missing value on or prior to Day 1. Population: Only participants with available data were analyzed.
  mg/dL
    number analyzed (Participants) | 86 | 180 | 266
    (all) | 115.8 (23.47) | 123.3 (26.48) | 120.9 (25.75)
High-sensitivity C-reactive protein (hsCRP) [Median (Full Range); unit: mg/dL] — Baseline was defined as the last non-missing value on or prior to Day 1. Population: Only participants with available data were analyzed.
  mg/dL
    number analyzed (Participants) | 86 | 180 | 266
    (all) | 2.260 [0.13 to 14.37] | 2.205 [0.22 to 39.20] | 2.215 [0.13 to 39.20]
Triglycerides (TGs) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the last two non-missing values on or prior to Day 1.
  mg/dL | 143.39 (61.932) | 166.93 (75.683) | 159.23 (72.213)
High-density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] — Baseline was defined as the mean of the last two non-missing values on or prior to Day 1.
  mg/dL | 57.07 (21.319) | 55.84 (16.326) | 56.24 (18.080)
Systolic blood pressure [Mean (Standard Deviation); unit: millimeter of mercury (mmHg)] | 126.0 (13.50) | 127.3 (13.34) | 126.9 (13.38)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 77.0 (7.56) | 76.4 (8.46) | 76.6 (8.17)
Body mass index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m2)] | 30.45 (5.787) | 29.52 (4.740) | 29.83 (5.114)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 12 in Low-Density Lipoprotein Cholesterol (LDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: ([LDL-C value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100. Bempedoic Acid = BA. Percent change from Baseline in LDL-C was analyzed using an analysis of covariance (ANCOVA) model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate. In the ANCOVA model, missing LDL-C data at Week 12 were imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Week 12
Population: Full Analysis Set: all randomized participants
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
percent change | 4.99 (2.299) | -23.46 (1.945)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -28.45, 95% CI 2-sided [-34.376 to -22.531], Standard Error of Mean 3.022

2. Secondary Outcome: Percent Change From Baseline to Week 12 in Non-high-density Lipoprotein Cholesterol (Non-HDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analysed for non-HDL-C. Baseline was defined as the mean of the non-HDL-C values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: ([non-HDL-C value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100. Percent change from Baseline in non-HDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate. In the ANCOVA model, missing non-HDL-C data at Week 12 were imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
percent change | 5.19 (2.202) | -18.38 (1.668)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -23.56, 95% CI 2-sided [-29.005 to -18.121], Standard Error of Mean 2.777

3. Secondary Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol (TC)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analysed for TC. Baseline was defined as the mean of the TC values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: ([TC value at Week 12 minus Baseline value] divided by [Baseline Value]) multiplied by 100. Percent change from Baseline in TC was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate. In the ANCOVA model, missing TC data at Week 12 were imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
Percent change | 2.88 (1.553) | -15.11 (1.282)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -17.99, 95% CI 2-sided [-21.940 to -14.030], Standard Error of Mean 2.018

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Apolipoprotein B (apoB)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analysed for apoB. Baseline was defined as the last non-missing value on or prior to Day 1. Percent change from baseline was calculated as: [(apoB value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Percent change from Baseline in apoB was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate. In the ANCOVA model, missing apoB data at Week 12 were imputed using multiple imputation method taking into account adherence to treatment.
Time Frame: Week 12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
Percent change | 4.74 (1.786) | -14.58 (1.497)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -19.32, 95% CI 2-sided [-23.908 to -14.732], Standard Error of Mean 2.341

5. Secondary Outcome: Percent Change From Baseline to Week 12 in High-sensitivity C-reactive Protein (hsCRP)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analysed for hsCRP. Baseline was defined as the last non-missing value on or prior to Day 1. Percent change from baseline was calculated as: [(hsCRP value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100.
Time Frame: Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 81 | 175
Percent change | 2.088 [-32.143 to 49.224] | -32.521 [-55.556 to 10.714]
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p < 0.001, Wilcoxon Rank Sum Test; Location shift = -31.045, 95% CI 2-sided [-44.761 to -17.401] — The location shift and asymptotic 95% confidence interval are based on Hodges-Lehman estimation

6. Secondary Outcome: Percent Change From Baseline to Week 12 in Triglycerides (TGs)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for TGs. Baseline was defined as the mean of the TGs values from the last two non-missing values on or prior to D 1. Percent change from baseline was calculated as: [(TGs value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Percent change from Baseline in TGs was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate.
Time Frame: Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 82 | 176
Percent change | 9.23 (4.218) | 4.70 (3.068)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p = 0.388, ANCOVA; Difference in LS mean = -4.53, 95% CI 2-sided [-14.877 to 5.812], Standard Error of Mean 5.240

7. Secondary Outcome: Percent Change From Baseline to Week 12 in High-density Lipoprotein Cholesterol (HDL-C)
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for HDL-C. Baseline was defined as the mean of the HDL-C values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: [(HDL-C value at Week 12 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Percent change from Baseline in HDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate.
Time Frame: Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 82 | 175
percent change | -1.38 (1.389) | -7.27 (1.214)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Test type: Superiority; p = 0.002, ANCOVA; Difference in LS mean = -5.89, 95% CI 2-sided [-9.528 to -2.250], Standard Error of Mean 1.845

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs, defined as an adverse events (AEs) that began or worsened in severity after the first dose of double-blind study drug and prior to the last dose of double-blind study drug + 30 days, were collected and reported.
Time Frame: Up to approximately 16 weeks
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study medication. Participants were included in the treatment group that they actually received, regardless of their randomized treatment.
Measure: Number; unit: Participants
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 87 | 181
Participants
  TEAEs | 39 | 88
  Non-serious TEAEs | 18 | 46
  Serious TEAEs | 3 | 5
  Deaths | 0 | 0

9. Other Pre Specified Outcome: Percent Change From Baseline to Weeks 4 and 8 in LDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for LDL-C. Baseline was defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: [(LDL-C value at Week 4 or 8 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Percent change from Baseline in LDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate.
Time Frame: Week 4 and Week 8
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
Percent change
  Week 4: number analyzed (Participants) | 85 | 180
  Week 4 | 3.05 (1.442) | -28.04 (1.704)
  Week 8: number analyzed (Participants) | 82 | 173
  Week 8 | 3.61 (1.773) | -25.51 (1.773)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -31.09, 95% CI 2-sided [-35.498 to -26.682], Standard Error of Mean 2.238
Statistical Analysis 2: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 8; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -29.12, 95% CI 2-sided [-34.074 to -24.168], Standard Error of Mean 2.513

10. Other Pre Specified Outcome: Percent Change From Baseline to Weeks 4 and 8 in Non-HDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for Non-HDL-C. Baseline was defined as the mean of the Non-HDL-C values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: [(Non-HDL-C value at Week 4 or 8 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Percent change from Baseline in non-HDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate.
Time Frame: Week 4 and Week 8
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
Percent change
  Week 4: number analyzed (Participants) | 85 | 180
  Week 4 | 3.08 (1.362) | -22.17 (1.457)
  Week 8: number analyzed (Participants) | 82 | 173
  Week 8 | 3.71 (1.660) | -20.04 (1.531)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -25.26, 95% CI 2-sided [-29.204 to -21.308], Standard Error of Mean 2.004
Statistical Analysis 2: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 8; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -23.75, 95% CI 2-sided [-28.219 to -19.276], Standard Error of Mean 2.268

11. Other Pre Specified Outcome: Percent Change From Baseline to Weeks 4 and 8 in TC
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analyzed for TC. Baseline was defined as the mean of the TC values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: [(TC value at Week 4 or 8 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Percent change from Baseline in TC was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate.
Time Frame: Week 4 and Week 8
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
Percent change
  Week 4: number analyzed (Participants) | 85 | 180
  Week 4 | 2.08 (1.000) | -18.33 (1.129)
  Week 8: number analyzed (Participants) | 82 | 173
  Week 8 | 1.82 (1.110) | -16.63 (1.215)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -20.41, 95% CI 2-sided [-23.390 to -17.430], Standard Error of Mean 1.513
Statistical Analysis 2: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 8; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -18.46, 95% CI 2-sided [-21.710 to -15.206], Standard Error of Mean 1.651

12. Other Pre Specified Outcome: Percent Change From Baseline to Weeks 4 and 8 in TGs
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analysed for TGs. Baseline was defined as the mean of the TGs values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: [(TGs value at Week 4 or 8 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Percent change from Baseline in TGs was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate.
Time Frame: Week 4 and Week 8
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
Percent change
  Week 4: number analyzed (Participants) | 85 | 180
  Week 4 | 6.00 (4.273) | 5.20 (2.536)
  Week 8: number analyzed (Participants) | 82 | 173
  Week 8 | 7.68 (4.246) | 7.60 (2.849)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 4; Test type: Superiority; p = 0.873, ANCOVA; Difference in LS mean = -0.8, 95% CI 2-sided [-10.663 to 9.059], Standard Error of Mean 4.990
Statistical Analysis 2: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 8; Test type: Superiority; p = 0.988, ANCOVA; Difference in LS mean = -0.08, 95% CI 2-sided [-10.215 to 10.055], Standard Error of Mean 5.131

13. Other Pre Specified Outcome: Percent Change From Baseline to Weeks 4 and 8 in HDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analysed for HDL-C. Baseline was defined as the mean of the HDL-C values from the last two non-missing values on or prior to Day 1. Percent change from baseline was calculated as: [(HDL-C value at Week 4 or 8 minus Baseline value) divided by (Baseline Value)] multiplied by 100. Percent change from Baseline in HDL-C was analyzed using an ANCOVA model with percent change from Baseline as the dependent variable, treatment as a fixed effects and Baseline as a covariate.
Time Frame: Week 4 and Week 8
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
Percent change
  Week 4: number analyzed (Participants) | 85 | 180
  Week 4 | 0.85 (1.204) | -7.73 (1.081)
  Week 8: number analyzed (Participants) | 82 | 173
  Week 8 | -1.33 (1.272) | -7.75 (1.144)
Statistical Analysis 1: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 4; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -8.59, 95% CI 2-sided [-11.778 to -5.394], Standard Error of Mean 1.619
Statistical Analysis 2: Comparison: Placebo vs Bempedoic Acid; Change from Baseline to Week 8; Test type: Superiority; p < 0.001, ANCOVA; Difference in LS mean = -6.42, 95% CI 2-sided [-9.798 to -3.049], Standard Error of Mean 1.712

14. Other Pre Specified Outcome: Absolute Change From Baseline to Weeks 4, 8, and 12 in LDL-C
Description: Blood samples were drawn after a minimum 10-hour fast (water was allowed) at pre-specified intervals. Samples were collected and analysed for LDL-C. Baseline was defined as the mean of the LDL-C values from the last two non-missing values on or prior to Day 1. Absolute change from baseline was calculated as: LDL-C value at Week 4, 8, or 12 minus Baseline value.
Time Frame: Week 4, Week 8 and Week 12
Population: Full Analysis Set. Only participants with available data were analyzed.
Measure: Geometric Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Bempedoic Acid
Number analyzed (Participants) | 88 | 181
milligrams per deciliter (mg/dL)
  Change from Baseline at Week 4: number analyzed (Participants) | 85 | 180
  Change from Baseline at Week 4 | 3.6 (15.65) | -37.4 (30.90)
  Change from Baseline at Week 8: number analyzed (Participants) | 82 | 173
  Change from Baseline at Week 8 | 3.9 (19.22) | -34.5 (32.29)
  Change from Baseline at Week 12: number analyzed (Participants) | 82 | 175
  Change from Baseline at Week 12 | 5.3 (23.96) | -32.9 (34.14)

ADVERSE EVENTS:
Time Frame: Up to approximately 16 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as an adverse events (AEs) that began or worsened in severity after the first dose of double-blind study drug and prior to the last dose of double-blind study drug + 30 days, were collected and reported. The analysis was performed using the Safety Analysis Set.
Arm/Group | Placebo | Bempedoic Acid
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/181
Serious Adverse Events (participants affected / at risk) | 3/87 | 5/181
Other Adverse Events (participants affected / at risk) | 18/87 | 46/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | Bempedoic Acid (N=181)
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Poisoning deliberate (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | Bempedoic Acid (N=181)
Vertigo (Ear and labyrinth disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 5
Nasopharyngitis (Infections and infestations) | 1 | 4
Urinary tract infection (Infections and infestations) | 5 | 5
Sinusitis (Infections and infestations) | 0 | 5
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0
Blood uric acid increase (Investigations) | 2 | 14
Liver function test increased (Investigations) | 0 | 7
Glomerular filtration rate decreased (Investigations) | 0 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 6
Headache (Nervous system disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT03001076/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/76/NCT03001076/SAP_001.pdf